CLINICAL TRIAL: NCT05354154
Title: Incidence of Postoperative Sore Throat and Risks Analysis in Patients Undergoing General Anesthesia With Endotracheal Intubation: A Prospective Cross-sectional Study
Brief Title: Incidence of Postoperative Sore-throat Incidence
Acronym: InciPost
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rehman Medical Institute - RMI (Other)
Responsible Party: Principal Investigator, Mohammad Shafiq, Principal investigator, Rehman Medical Institute - RMI
Other Study IDs: RMI/RMI-REC/Approval/126
Record Dates: First submitted 2022-04-25; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Sore-throat
MeSH Terms: conditions — Pharyngitis | interventions — Intubation, Intratracheal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: endotracheal intubation — Consenting healthy patients of either sex will be endotracheally intubated under controlled environment

SUMMARY:
Postoperative sore throat is a distressing but frequent symptom presented by the patients on the floor upon awakening from General Anesthesia, where endotracheal intubation is part of the Anesthetic protocol. Its incidence ranges between 21-71.8%. Good skills and availability of trained staff to cause minimal tissue damage are expected to reduce the incidence. Risks factors associated will be analyzed.

DETAILED DESCRIPTION:
Post-operative sore throat (POST) is a common complication of endotracheal intubation. It ranges from 21 to 71.8 %. Various factors contribute to the development of POST, like, female sex, smoking, intubation difficulty and Suxamethonium use, high endotracheal cuff pressure, airway suctioning, long duration of surgery, mucosal injury with laryngoscopy, or pharyngeal airway use and larger size endotracheal tubes [9]. POST has also been associated with laryngeal masks, injury with laryngoscopy, or pharyngeal airway use and larger size endotracheal tubes. Basically it is mucosal damage of the throat and trachea which releases inflammatory mediators and produces soreness. POST leads to postoperative dissatisfaction. Patients of POST are uncontended following general anesthesia. Its preemptive amelioration, has been studied using various pharmacological interventions. The list includes, but is not limited to, Benzydamine hydrochloride (BH), aspirin, ketamine, lidocaine and dexamethasone. There is limited evidence based literature available about the incidence of POST in the investigator's locality in the country. The investigators plan to collect data in General OT of Rehman Medical institute (RMI), Peshawar. The city of Peshawar is the largest city of Khyber Pakhtunkhwa, a province of Pakistan, having a population of approximately 2 million. The objectives of our study is to know the magnitude of the problem and ascertain factors associated with postoperative sore throat among patients undergoing elective surgery under general anesthesia with endotracheal intubation.

ELIGIBILITY:
Inclusion Criteria:

* Any patient of either gender aged 18- 60 years
* Patients of American Society of Anesthesiologists (ASA) physical status 1 and 2 receiving General Anesthesia with ETT

Exclusion Criteria:

* Patients having ASA 3 or above physical status
* Recent or ongoing Upper Respiratory Tract Infection (URTI)
* Patients going to ICU intubated

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population is all inpatients admitted in surgical and allied departments.
Sampling Method: Probability Sample
Enrollment: 249 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of sorethroat | Six hours
  Incidence= Those who developed Postoperative sorethroat / All recruited participants who recieve General anesthesia through endotracheal tubes *100

SECONDARY OUTCOMES:
Risk factors assessment | Six hours
  Associated risk factors for postoperative Sore throat will be assessed for presence or absence through a structured performa

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Shafiq, FCPS, Principal Investigator — Rehman Medical Institute
Locations (1):
- Rehman Medical Institute, Peshawar, Khyber Pakhtunkhwa, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Data including clinical and demographic characteristics, not affecting patient's confidentiality, will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: April, 2022 to April, 2025
Access Criteria: IPD will be shared on inter institutional request basis.

REFERENCES:
- [Background] Gupta D, Agrawal S, Sharma JP. Evaluation of preoperative Strepsils lozenges on incidence of postextubation cough and sore throat in smokers undergoing anesthesia with endotracheal intubation. Saudi J Anaesth. 2014 Apr;8(2):244-8. doi: 10.4103/1658-354X.130737. PMID 24843341
- [Background] Alcock R, Peachey T, Lynch M, McEwan T. Comparison of alfentanil with suxamethonium in facilitating nasotracheal intubation in day-case anaesthesia. Br J Anaesth. 1993 Jan;70(1):34-7. doi: 10.1093/bja/70.1.34. PMID 8431329
- [Background] Joe HB, Kim DH, Chae YJ, Kim JY, Kang M, Park KS. The effect of cuff pressure on postoperative sore throat after Cobra perilaryngeal airway. J Anesth. 2012 Apr;26(2):225-9. doi: 10.1007/s00540-011-1293-2. Epub 2011 Nov 30. PMID 22127511
- [Background] Mencke T, Noeldge-Schomburg G. Laryngeal morbidity after use of the laryngeal mask airway. Acta Anaesthesiol Scand. 2010 Feb;54(2):127-8. doi: 10.1111/j.1399-6576.2009.02159.x. No abstract available. PMID 20078448
- [Background] Canbay O, Celebi N, Sahin A, Celiker V, Ozgen S, Aypar U. Ketamine gargle for attenuating postoperative sore throat. Br J Anaesth. 2008 Apr;100(4):490-3. doi: 10.1093/bja/aen023. Epub 2008 Mar 1. PMID 18310675
- [Background] Xu YJ, Wang SL, Ren Y, Zhu Y, Tan ZM. A smaller endotracheal tube combined with intravenous lidocaine decreases post-operative sore throat - a randomized controlled trial. Acta Anaesthesiol Scand. 2012 Nov;56(10):1314-20. doi: 10.1111/j.1399-6576.2012.02768.x. Epub 2012 Sep 24. PMID 22999067
- [Background] Patki A. Laryngeal mask airway vs the endotracheal tube in paediatric airway management: A meta-analysis of prospective randomised controlled trials. Indian J Anaesth. 2011 Sep;55(5):537-41. doi: 10.4103/0019-5049.89900. PMID 22174478
- [Background] Jaensson M, Gupta A, Nilsson UG. Risk factors for development of postoperative sore throat and hoarseness after endotracheal intubation in women: a secondary analysis. AANA J. 2012 Aug;80(4 Suppl):S67-73. PMID 23248834
- [Background] Bagchi D, Mandal MC, Das S, Sahoo T, Basu SR, Sarkar S. Efficacy of intravenous dexamethasone to reduce incidence of postoperative sore throat: A prospective randomized controlled trial. J Anaesthesiol Clin Pharmacol. 2012 Oct;28(4):477-80. doi: 10.4103/0970-9185.101920. PMID 23225928
- [Background] Chen CY, Kuo CJ, Lee YW, Lam F, Tam KW. Benzydamine hydrochloride on postoperative sore throat: a meta-analysis of randomized controlled trials. Can J Anaesth. 2014 Mar;61(3):220-8. doi: 10.1007/s12630-013-0080-y. Epub 2013 Nov 22. PMID 24263969
- [Background] Agarwal A, Nath SS, Goswami D, Gupta D, Dhiraaj S, Singh PK. An evaluation of the efficacy of aspirin and benzydamine hydrochloride gargle for attenuating postoperative sore throat: a prospective, randomized, single-blind study. Anesth Analg. 2006 Oct;103(4):1001-3. doi: 10.1213/01.ane.0000231637.28427.00. PMID 17000820
- [Background] Mayhood J, Cress K. Effectiveness of ketamine gargle in reducing postoperative sore throat in patients undergoing airway instrumentation: a systematic review. JBI Database System Rev Implement Rep. 2015 Sep;13(9):244-78. doi: 10.11124/jbisrir-2015-2045. PMID 26470672
- [Background] Tanaka Y, Nakayama T, Nishimori M, Tsujimura Y, Kawaguchi M, Sato Y. Lidocaine for preventing postoperative sore throat. Cochrane Database Syst Rev. 2015 Jul 14;2015(7):CD004081. doi: 10.1002/14651858.CD004081.pub3. PMID 26171894
- [Background] Kuriyama A, Maeda H. Preoperative intravenous dexamethasone prevents tracheal intubation-related sore throat in adult surgical patients: a systematic review and meta-analysis. Can J Anaesth. 2019 May;66(5):562-575. doi: 10.1007/s12630-018-01288-2. Epub 2019 Jan 7. PMID 30617677
- [Result] Lee JY, Sim WS, Kim ES, Lee SM, Kim DK, Na YR, Park D, Park HJ. Incidence and risk factors of postoperative sore throat after endotracheal intubation in Korean patients. J Int Med Res. 2017 Apr;45(2):744-752. doi: 10.1177/0300060516687227. Epub 2017 Feb 7. PMID 28173712
- [Result] Scuderi PE. Postoperative sore throat: more answers than questions. Anesth Analg. 2010 Oct;111(4):831-2. doi: 10.1213/ANE.0b013e3181ee85c7. No abstract available. PMID 20870978